CLINICAL TRIAL: NCT00514501
Title: Open-label, Phase 2 Study of the Safety and Efficacy of B-methyl-P-(123I)- Iodophenyl-pentadecanoic Acid (Iodofiltic Acid I 123) For Identification of Ischemic Myocardium Using Single Photon Emission Computed Tomography (Spect) in Adults With Symptoms Consistent With Acute Coronary Syndrome (ACS).
Brief Title: Safety and Efficacy Iodofiltic Acid I 123 in the Treatment of Acute Coronary Syndrome
Acronym: Zeus-ACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIP-BP23; NCT00585663 (obsolete NCT alias)
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — iodofiltic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iodofiltic Acid I 123 (Experimental)
  Interventions: Drug: Iodofiltic acid I 123

INTERVENTIONS:
Drug: Iodofiltic acid I 123

SUMMARY:
This is an open-label phase 2 study recruiting low, moderate, and high likelihood ACS patients from approximately 60 centers. Patients will be imaged with iodofiltic acid I 123 for the detection of myocardial ischemia. Readers independent of the clinical study centers will review results of imaging studies in a blinded fashion at an imaging core lab. The resulting independent reading of the images will be compared against the truth standard for ACS.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and are willing to comply with protocol requirements
* Are 40 years of age or older.
* Are being evaluated for possible ACS.
* If female, then not of childbearing potential as documented by history or has a negative serum or urine pregnancy test within 4 hours prior to receiving the test drug and agrees to use an acceptable form of birth control.

Exclusion Criteria:

* <40 years of age.
* Females who are pregnant or lactating.
* History of left ventricular ejection fraction (LVEF)=40%.
* History of MI.
* Acute ST segment elevation on ECG.
* Left bundle branch block on ECG.
* Known history of significant allergy to x-ray contrast media or iodine/iodides.
* Currently or formerly on medication that targets fatty acid uptake or metabolism, eg ranolazine, (Ranexa).
* Administered radiopharmaceutical other than rubidium-82 or thallium-201 within 2 days prior to study enrollment.
* Underwent cardiac stress testing of any kind within 2 days prior to study enrollment.
* Serum creatinine level >2.0 mg per dL.
* Received investigational compound and/or medical device within 30 days of admission into this study.
* Q-wave abnormalities consistent with previous MI

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman LaFrance, MD, Study Director — Molecular Insight Pharmaceuticals, Inc.
Locations (38):
- United States (36):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Los Angeles, California
  - Mission Viejo, California
  - Newport Beach, California
  - Roseville, California
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Newark, Delaware
  - Jacksonville, Florida
  - Aurora, Illinois
  - Maywood, Illinois
  - Louisville, Kentucky
  - Auburn, Maine
  - Bethesda, Maryland
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Manchester, New Hampshire
  - Albany, New York
  - Brooklyn, New York
  - Kingston, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Providence, Rhode Island
  - Houston, Texas
  - Richmond, Virginia
  - Madison, Wisconsin
- Canada (2):
  - North Vancouver, British Columbia
  - Scarborough Village, Ontario

REFERENCES:
- [Derived] Kontos MC, Dilsizian V, Weiland F, DePuey G, Mahmarian JJ, Iskandrian AE, Bateman TM, Heller GV, Ananthasubramaniam K, Li Y, Goldman JL, Armor T, Kacena KA, LaFrance ND, Garcia EV, Babich JW, Udelson JE. Iodofiltic acid I 123 (BMIPP) fatty acid imaging improves initial diagnosis in emergency department patients with suspected acute coronary syndromes: a multicenter trial. J Am Coll Cardiol. 2010 Jul 20;56(4):290-9. doi: 10.1016/j.jacc.2010.03.045. PMID 20633821

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodofiltic Acid I 123: A single IV dose of iodofiltic acid I 123 (approximately 4.0-5.0 mCi) was injected through an indwelling catheter, followed by 10 mL of normal saline to complete delivery of the dose.
Period: Overall Study
Arm/Group | Iodofiltic Acid I 123
Started | 510
Completed | 507
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Iodofiltic Acid I 123
Number analyzed (Participants) | 507
Age, Continuous [Mean (Full Range); unit: years] | 59.2 [30 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232
  Male | 275

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity of Detecting Myocardial Ischemia (Reader 1)
Description: Enrolled subjects were imaged (10 minutes post-injection) using iodofiltic acid I 123 SPECT and the resulting data were reviewed in blinded reads by readers independent of the study centers and the Sponsor. The results obtained in these blinded reads were compared with the final diagnosis for each subject with regard to myocardial ischemia or ACS, determined by the Final Diagnosis Clinical Endpoints Committee (FDCEC).
  Sensitivity = % (n/N): N = number of subjects positive for ischemia per the FDCEC; n = subset of N positive for ischemia per the blinded Majority Read (two of three readers) of iodofiltic acid I 123 readers.
  Specificity = % (n/N): N = number of subjects negative for ischemia per the FDCEC; n = subset of N negative for ischemia per the blinded Majority Read (two of three readers) of iodofiltic acid I 123 readers.
Time Frame: Day 30
Population: The study enrolled a total of 510 subjects; 507 of these subjects received iodofiltic acid I 123, and 506 had iodofiltic acid I 123 SPECT images available. Of the 507 subjects who were dosed, 342 were eligible for efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: % (n/N)
Arm/Group | Iodofiltic Acid I 123
Number analyzed (Participants) | 342
% (n/N)
  Sensitivity | 75.2 [66.8 to 83.6]
  Specificity | 67.7 [61.4 to 74.0]

2. Primary Outcome: Sensitivity, Specificity of Detecting Myocardial Ischemia (Reader 2)
Description: as for outcome 1
Time Frame: Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % (n/N)
Arm/Group | Iodofiltic Acid I 123
Number analyzed (Participants) | 342
% (n/N)
  Sensitivity | 75.2 [66.8 to 83.6]
  Specificity | 59.8 [53.3 to 66.4]

3. Primary Outcome: Sensitivity, Specificity of Detecting Myocardial Ischemia (Reader 3)
Description: as for outcome 1
Time Frame: Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % (n/N)
Arm/Group | Iodofiltic Acid I 123
Number analyzed (Participants) | 342
% (n/N)
  Sensitivity | 74.3 [65.8 to 82.8]
  Specificity | 71.6 [65.6 to 77.7]

ADVERSE EVENTS:
Arm/Group | Iodofiltic Acid I 123
Serious Adverse Events (participants affected / at risk) | 28/507
Other Adverse Events (participants affected / at risk) | 32/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodofiltic Acid I 123 (N=507)
Cardiac failure, acute (Cardiac disorders) | 2 (3)
Cardiac arrest (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mental status changes (Nervous system disorders) | 1 (1)
Chest pain (Cardiac disorders) | 4 (5)
Myocardial infarction (Cardiac disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Unstable angina (Cardiac disorders) | 3 (3)
Aortic dissection (Cardiac disorders) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodofiltic Acid I 123 (N=507)
Dysgeusia (Nervous system disorders) | 12 (12)
Headache (Nervous system disorders) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less